CLINICAL TRIAL: NCT04320433
Title: Inter-day Reliability of the Oral Glucose Tolerance Test Using Indirect Calorimetry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Associate professor, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1102/CEIH/2020
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Participants will undergo two trials visit (with a week of separation). During the visits they will ingest an oral glucose load solution (oral glucose tolerance test) and gas exchange will be measured over the following 3-hours. The glucose levels will be monitored through a Glucose meter in different time frames.
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — Participants will ingest 75g anhydrous glucose dissolved in a volume of 200mL of water (NUTER.TEC GLUCOS, Subra, Toulouse, France).

SUMMARY:
The main aim of this study is to determine the inter-day reliability, by using indirect calorimetry, of the post-prandial macronutrient oxidation and energy expenditure after consuming oral glucose load solution.

DETAILED DESCRIPTION:
The maintenance of blood glucose concentrations and the oxidation of carbohydrate after consuming carbohydrate is related with a low risk of mortality and morbidity from cardiometabolic diseases. The oral glucose tolerance test is a diagnostic test widely used in the clinical field. However, its inter-day reliability has not been deeply studied. Therefore, it is of clinical interest to study the inter-day reliability of the diagnostic test oral glucose tolerance test using indirect calorimetry and monitoring the response of the glucose levels.

20 young adults will undergo two trials visit with 7 days of separation between conditions. Each evaluation day will conform to the following tests:

1. Basal metabolic rate assessment through indirect calorimetry.
2. Basal heart rate variability through heart rate monitor.
3. Intake of the corresponding glucose load solution.
4. Postprandial nutrient oxidation and energy expenditure assessment through indirect calorimetry
5. Glucose monitoring through Glucose meter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Ages 18-30 years
* BMI: 18-27.5 kg/m2
* Stable weight over the last 3 months (body weight changes<35kg)
* Participant must be capable and willing to provide consent, understand exclusion criteria, instructions and protocols.

Exclusion Criteria:

* History of cardiovascular disease
* Diabetes or hypertension
* Pregnant, planning to become pregnant, or breastfeeding
* Have been treated previously or during the study period with prescription drugs: antihypertensive, lipid lowering, acid uric lowering, glucose lowering, beta blockers or any drug that under the investigator's judged could influence the results.
* Any non-controlled medical condition which could influence results or could be worsened by the participation in the study.
* Claustrophobia
* Needle phobia
* Are deemed unsuitable by the investigator for any other reason, that prevent data collection.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Inter-day reliability, 7 days apart, in post-prandial nutrient oxidation | 7 days
  Reliability

SECONDARY OUTCOMES:
Inter-day reliability, 7 days apart, in post-prandial energy expenditure | 7 days
  Reliability
Inter-day reliability, 7 days apart, in glucose levels | 7 days
  Reliability

OTHER OUTCOMES:
• Reliability of the O2 and CO2 metabolic cart sensors by pure gases infusions using a high-precision mass-flow controllers | Immediately after the participants' gas exhange measurements
  o Inter-day reliability of gas composition (O2 and CO2) measurement by the Omnical® assessed by comparison with a high-precision mass-flow controllers.

CONTACTS AND LOCATIONS:
Overall Officials: juanma.alcantara@hotmail.com Ruiz Ruiz, Dr., Principal Investigator — Universidad de Granada
Locations (1):
- Jonatan Ruiz Ruiz, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alcantara JMA, Sanchez-Delgado G, Jurado-Fasoli L, Galgani JE, Labayen I, Ruiz JR. Reproducibility of the energy metabolism response to an oral glucose tolerance test: influence of a postcalorimetric correction procedure. Eur J Nutr. 2023 Feb;62(1):351-361. doi: 10.1007/s00394-022-02986-w. Epub 2022 Aug 25. PMID 36006468